CLINICAL TRIAL: NCT03549182
Title: The Influence of Acute Tryptophan Depletion on Emotion and Interference Processing and Potential Moderation by 5HT Genetics (TPH2)
Brief Title: Serotonin, Serotonin Genetics(TPH2) and Emotion and Interference Processing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Benjamin Becker, Professor, University of Electronic Science and Technology of China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: UESTC-neuSCAN-51
Record Dates: First submitted 2018-02-05; First posted 2018-06-07 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Healthy
Keywords: acute tryptophan depletion; tryptophan hydroxylase 2 gene; emotion

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- male TPH2-GG carriers with ATD then placebo group (Experimental): male TPH2-GG carriers will first receive ATD, then will receive placebo at least 5 weeks later.
  Interventions: Drug: ATD treatment; Drug: placebo treatment
- male TPH2-GG carriers with placebo then ATD group (Experimental): male TPH2-GG carriers will first receive placebo, then will receive ATD at least 5 weeks later.
  Interventions: Drug: ATD treatment; Drug: placebo treatment
- male TPH2-TTcarriers with ATD then placebo group (Experimental): male TPH2-TT carriers will first receive ATD, then will receive placebo at least 5 weeks later.
  Interventions: Drug: ATD treatment; Drug: placebo treatment
- male TPH2-TTcarriers with placebo then ATD group (Experimental): male TPH2-TT carriers will first receive placebo,then will receive ATD at least 5 weeks later.
  Interventions: Drug: ATD treatment; Drug: placebo treatment

INTERVENTIONS:
Drug: ATD treatment — oral administration of ATD (100g)(Acute Tryptophan Depletion)
Drug: placebo treatment — oral administration of placebo (102.3g)

SUMMARY:
The study aims to explore whether acute tryptophan depletion can affect the emotion and interference processing whether this effect is moderated by the TPH2 genotype

DETAILED DESCRIPTION:
Based on previous studies suggesting that serotonin, a neurotransmitter, is associated with social & emotional behavior, including emotional reactivity and emotion regulation, the present study aims to explore effects of acute tryptophan depletion (ATD) on emotion processing and emotional interference processing within a randomized double-blind, with-subject, placebo-controlled pharmaco-fMRI experiment. To further examine the potential moderating effects of the genetic makeup of the serotonin system the present study will include a pharmacogenetics imaging approach. Given that TPH2 is the key regulator of the serotonergic signaling pathway, we therefore assessed whether such the effects of tryptophan depletion vary according to the TPH2 genotype. To this end, healthy male TPH2-GG or TPH2-TT carriers will be recruited and will receive ATD (100g) and placebo (102.3g) in a within subject design. To control for potential effects of pre-medication personality traits as well as effects of medicines on mood, subjects will be administered pre-treatment assessing relevant personality traits and post-treatment assessments of mood.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects without past or current psychiatric or neurological disorders
* Right-handedness

Exclusion Criteria:

* History of head injury;
* Medical or psychiatric illness.
* High blood pressure, general cardio-vascular alterations
* History of drug or alcohol abuse or addiction.
* Allergy against medications or general strong allergies
* Sleep disorders.
* Visual or motor impairments

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Neural processing during emotion processing as assessed via fMRI | 5-6h after administration of ATD, or placebo
  Subjects will undergo a validated emotional face paradigm. To assess genotype x ATD interaction effects on neural emotional reactivity effects of ATD depletion on the corresponding neural activity will be compared between the TPH2 genotype groups.
Neural processing during interference processing as assessed via fMRI | 5-6h after administration of ATD, or placebo
  Subjects will undergo a validated cognitive-emotional interference paradigm. To assess genotype x ATD interaction effects on neural interference control effects of ATD depletion on the corresponding neural activity will be compared between the TPH2 genotype groups.
Neural processing during the resting state as assessed via fMRI | 5-6h after administration of ATD, or placebo
  Subjects will undergo a validated resting state assessment. To assess genotype x ATD interaction effects on intrinsic brain activity in the emotion and interreference related neural networks effects of ATD depletion on the corresponding neural activity will be compared between the TPH2 genotype groups.

SECONDARY OUTCOMES:
Behavioral interference performance | 5-6h after administration of ATD, or placebo
  Subjects will undergo a emotion-cognition interference paradigm. To assess genotype x ATD interaction effects on behavioral indices of interference (congruent vs incongruent trials) behavioral performance (accuracy/reaction time) effects of ATD depletion on the corresponding behavioral indices will be compared between the TPH2 genotype groups.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Life Science and Technology, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No